### CLINICAL TRIAL PROTOCOL

# ASSESSMENT OF THE INCREMENTAL HAEMODIALYSIS SECURITY AND EFFECTIVENESS IN INCIDENT PATIENTS

PROTOCOL CODE

Trial IHDIP

**VERSION:** 

2nd version of March 10th 2017

## SPONSOR and COORDINATOR/INVESTIGATORS:

Dr. Javier L. Deira Lorenzo Dr. Miguel A. Suárez Santisteban

Nephrology Department Nephrology Unit

Hospital Complex from Cáceres Hospital Virgen del Puerto from Plasencia

This project has the endorsement of the Extremadura Health and Social Policy Council and also of the Spanish Society of Nephrology





This document belongs to the sponsor and contains confidential information under professional secret. Neither this document, nor the information contained can be divulged, published, revealed or transferred in any way to a third person, in any form without the written consent from sponsor, with the exception of the Health Authorities and Ethical Committee that require it.

# **IINFORMED CONSENT**

| Hemodialysis modality: | |
|---|---|
| Progressive hemodialysis | |
| Conventional hemodialysis | |
| 1. Hospital: | |
| 2. Service/Unit | |
| 3. Doctor: | |
| 4. Patient: | |
| 5. ID: | |
| 6. Representative: | |
| 7. ID: | |
| The document is intended to verify that you, or whoever represents you, have received verl writing) adequate and understandable information, including the purpose and nature of procedure, its risks and consequences. As with any action in the field of health, for the accomposed of Hemodialysis (Progressive or Conventional) also requires the free and voluntary consequent, once all the information has been received and evaluation according to nat international regulation have been carried out. | the above<br>plishment<br>ent of the |
| I DECLARE: That the Doctor | nderstood<br>en able to<br>y consent,<br>ned of the<br>essing and<br>modialysis |
| In <i>(place)</i> del 201 | |
| Signed<br>Miss/Mrs/Mr/MsID | |

### ADDITIONAL INFORMATION ATTACHED TO THIS CONSENT

Your doctor has diagnosed you with a condition called advanced chronic kidney disease. Irreversibly, your kidneys do not perform their function effectively and as a result do not purify the blood of substances that are dangerous to life, nor are there other ones that are essential. Therefore, it is not possible to live without an organ that develops all these important functions. For this reason, his nephrologist believes that he must initiate a treatment that is known as hemodialysis (HD), which tries to supply, but only partially, some of the functions of his kidneys.

Dialysis consists of cleaning the blood, allowing the passage of water and substances contained in it, through a specific filter, which we call the dialyser, made a liquid for its elimination. This results in prolonged survival, which depends to a great extent on the age and associated diseases of the patients. Hemodialysis is usually well tolerated although occasional side effects may occur. Some common but not very serious:

- 1. Nausea, vomiting, headache, hypotension, cramps.
- 2. Hematomas or small blood loss from the puncture points or from a breakdown of the dialyzer.
- 3. Other uncommon but more serious as cardiac abnormalities such as arrhythmias, angina pectoris, or strokes, severe allergic reactions, or rupture of red blood cells (hemolysis). The latter could endanger your life in a very exceptional way.
- 4. In some cases, infectious complications may occur, due to the reduction of the hemodialysis patient's defenses, or to the manipulation of blood, and to the patient's contact in hospital settings. They are usually due to bacteria or viruses, and can cause hepatitis B and C.
- 5. There are other complications related to vascular access that occur in the form of hemorrhages, thrombosis, infections and, exceptionally, their rupture, involving medical rescue techniques and procedures.

As for the number of sessions per week of the same, we can say that their number is one that allows to improve the quality of life of the patient with the renal replacement technique. For this, several clinical guidelines recommend, based on the evidence, the dose and frequency of sessions. The KDOQI1 (International Hemodialysis Guide) recommends a minimum dose, measured by Kt / V of 1.2 for patients prevalent in the 3-week anuric session mode, but opens the door to adjust it conditioned to the existence or non-existence of function Renal residual. That is, if you urinate more than 500 milliliters a day and the elimination of toxins from your kidneys is higher than 2.5 ml / min, measured by your reference nephrologist (according to validated formulas), is a candidate, if there are no diseases that contraindicate to enter a HD session a week, unlike the usual pattern of 3 sessions. We rely on promising studies, which emphasize that starting hemodialysis once or twice a week versus three times a week, preserves residual renal function, with no associated complications. Furthermore, this residual renal function has been correlated with a decrease in morbidity and mortality in patients on dialysis programs. The possible complications, added to the previous ones are the possibility of VOLUME OVERLOAD OR A BAD CONTROL OF THE BASE-ACID BALANCE AND / OR THE HYPERPOTASEMIA. For this reason, it is important to monitor the patient's weight gain and the ultrafiltration rates necessary for maintenance. As well as necessary biochemical and gasometric controls (fortnightly or earlier) if a possible complication is suspected.

You have also been informed of your right to request additional information in case you need it, and that no additional procedure, other than those of which you have been informed, is given to you, for which you have given your consent, unless it is strictly necessary to save your life or to avoid some irreparable damage to your health. Finally, in compliance with the Law on the protection of personal data (*check national regulations*) we inform you that the information obtained in the healthcare of your person has been incorporated for treatment to an automated file. It is also informed that the collection

and treatment of these data are aimed at the epidemiological, scientific and educational study, respecting at all times their anonymity. If you wish, you can exercise the rights of access, rectification, cancellation and opposition, provided by law.

#